CLINICAL TRIAL: NCT00608153
Title: Compliance of Patients With Essential Hypertension Treated With Candesartan or Candesartan/Hydrochlorothiazide
Acronym: CoCa
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Andrea Pahor, AstraZeneca Germany
Other Study IDs: NIS-CGE-ATA-2007/1
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-01

CONDITIONS: Essential Hypertension
Keywords: essential hypertension; ARB; compliance; candesartan
MeSH Terms: conditions — Essential Hypertension; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patient with essential hypertension under treatment with candesartan or candesartan HCT

SUMMARY:
The CoCa study with at maximum daily dose of 32 mg candesartan or 16/12.5 mg candesartan/hydrochlorothiazide has the objective to evaluate under naturalistic conditions, i.e. under routine medical care conditions, the subject compliance as well as the efficacy and tolerability of candesartan or candesartan/HCT in subjects suffering from essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension
* under candesartan treatment

Exclusion Criteria:

-

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care ambulant patient
Sampling Method: Probability Sample
Enrollment: 1773 (Actual)
Dates: Start 2007-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To estimate under naturalistic conditions the compliance rate, defined as the number of subjects with regular intake of the prescribed dose of candesartan or candesartan/HCT as judged by the physician at the end of the observational period. | app. 3 monthly

SECONDARY OUTCOMES:
To assess under naturalistic conditions the subject's reason(s) for being compliant or non-compliant with the intake of the pre-scribed dose of candesartan or candesartan/HCT | app. 3 monthly
To assess under naturalistic conditions the subject's reason(s) for withdrawal of the pre-scribed dose of candesartan or candesartan/HCT | app. 3 monthly
To assess under naturalistic conditions whether physicians are using procedures to improve the subject's compliance regarding the intake of candesartan or candesartan/HCT and to get insight in the type and effects of these procedures | app. 3 monthly

CONTACTS AND LOCATIONS:
Overall Officials: R. E. Schmieder, MD, Principal Investigator — University hospital Erlangen-Nurnberg; Andrea Pahor, MD, Study Chair — MED Dep., AstraZeneca Germany